CLINICAL TRIAL: NCT02160249
Title: RISE (Rehabilitation Intervention for People With Schizophrenia in Ethiopia): a Cluster-randomised Trial
Brief Title: RISE (Rehabilitation Intervention for People With Schizophrenia in Ethiopia)
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Addis Ababa University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 7035; 100142/Z/12/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia Spectrum Disorder; Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Psychotic disorders; Schizophrenia spectrum disorder (schizophrenia, schizoaffective disorder or schizophreniform disorder) using DSM-IV criteria
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community-based rehabilitation and facility based care (Experimental): Community-based rehabilitation is delivered to participants and their caregivers at their home by a specialist CBR worker. It comprises psychoeducation, adherence support, rehabilitation (including self-care and social skills), family support groups and accessing existing community organisations. It also involves community awareness raising and education and mobilisation of community leaders.
  Facility based care (usual care) consists of anti-psychotic medication prescribed by a nurse or clinical officer in a health centre and basic psycho-education.
  Interventions: Behavioral: Community-based rehabilitation; Other: Facility based care
- Facility-based care (Active Comparator): Facility based care (usual care) consists of anti-psychotic medication prescribed by a nurse or clinical officer in a health centre and basic psycho-education.
  Interventions: Other: Facility based care

INTERVENTIONS:
Behavioral: Community-based rehabilitation
  Arms: Community-based rehabilitation and facility based care
Other: Facility based care

SUMMARY:
The purpose of this study is to determine whether community-based rehabilitation plus facility-based care is superior to facility-based care alone in reducing disability related to schizophrenia in rural Ethiopia.

DETAILED DESCRIPTION:
This is a cluster randomised trial set in rural Ethiopia with kebeles (villages) as the unit of randomisation. 54 kebeles will be included. 27 will be randomly allocated to the intervention arm (Facility based care (FBC) + Community-based Rehabilitation (CBR)) and 27 randomly allocated to the control arm (FBC alone).

The aim is to determine whether CBR + FBC is superior to FBC alone in reducing disability related to schizophrenia, measured by the WHO Disability Assessment Schedule version 2.0 (WHODAS 2.0) at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of schizophrenia spectrum disorder (schizophrenia, schizoaffective disorder or schizophreniform disorder) using (DSM-IV) criteria
* Evidence of severe, enduring or disabling illness
* Resident in kebele for >6 months and no immediate plans to leave the kebele
* Has a primary caregiver who is willing to participate in the study

Exclusion Criteria:

* No specific criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03-26 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Disability (36-item WHODAS (World Health Organisation Disability Assessment Schedule) 2.0) | 12 months

SECONDARY OUTCOMES:
Symptom severity (Brief Psychiatric Rating Scale- Expanded version (BPRS-E)) | 6 and 12 months
Clinical Global Impression (CGI) | 6 and 12 months
Relapse (Longitudinal Interval Follow up Evaluation: DSM-IV version (LIFE)) | 6 and 12 months
Disability (36-item WHODAS 2.0) | 6 months
Functioning (indigenous functioning scale) | 6 and 12 months
  Scale is currently under development. It is being designed and validated to measure functioning in people with severe mental illness in rural Ethiopia.
Economic activity of patient (employment, income and household work) | 6 and 12 months
  Section includes current occupation (categories), employment status (categories), typical income (specific amount). Section also includes questions adapted from the WHO-DAS 12 and 36 relating to problems doing usual work task both generally and as a result of their mental illness (likert scale)
Medication adherence (4 item Morisky Medication Adherence Scale) | 6 and 12 months
Engagement with facility based care | 6 and 12 months
  Potential mediator
Proportion with human rights problems (chaining or restraint)- self-reported | 6 and 12 months
  The outcome is the proportion chained, restrained or confined within last one month. Additional data on who perpetrated the chaining i.e. traditional healer/ family member will be collected.
Nutritional status (BMI) | 6 and 12 months
Serious adverse events | 6 and 12 months
Economic activity of caregiver | 6 and 12 months
  Section includes current occupation (categories), employment status (categories), typical income (specific amount). Section also includes questions adapted from the WHO-DAS 12 and 36 relating to problems doing usual work tasks (likert scale).
Caregiver burden (WHO Family Interview Schedule Impact section) | 6 and 12 months
Caregiver depression (PHQ9 +1) | 6 and 12 months
Patient medication adherence | 6 and 12 months
Proportion with human rights problems (chaining or restraint)- Caregiver-reported | 6 and 12 months
  Caregiver to report presence of human rights problems relating to patient. The outcome is the proportion chained, restrained or confined within last one month. Additional data on who perpetrated the chaining i.e. traditional healer/ family member will be collected.

OTHER OUTCOMES:
Discrimination (DISC-12) | 6 and 12 months
  Potential mediator
Health service use and costs | 6 and 12 months
  Potential mediator
Depression (PHQ-9+1) | 6 and 12 months
  Potential confounder
Access/ adherence to CBR and reasons for non-adherence | 6 and 12 months
  Potential mediator
Social support (OSLO-3) | 6 and 12 months
  Potential mediator
Stigma and discrimination (WHO Family Interview Schedule Stigma section) | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary De Silva, PhD MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Abebaw Fekadu, Principal Investigator — Addis Ababa University Department of Psychiatry
Locations (1):
- Department of Psychiatry, College of Health Sciences, Addis Ababa University, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Dijkstra LG, Weiss HA, Birhane R, Medhin G, de Silva M, Hanlon C, Fekadu A, Asher L. Effects of community-based rehabilitation on caregivers of people with schizophrenia in Ethiopia in the RISE trial. BMC Psychiatry. 2025 Mar 11;25(1):231. doi: 10.1186/s12888-025-06651-4. PMID 40069613
- [Derived] Asher L, Birhane R, Weiss HA, Medhin G, Selamu M, Patel V, De Silva M, Hanlon C, Fekadu A. Community-based rehabilitation intervention for people with schizophrenia in Ethiopia (RISE): results of a 12-month cluster-randomised controlled trial. Lancet Glob Health. 2022 Apr;10(4):e530-e542. doi: 10.1016/S2214-109X(22)00027-4. PMID 35303462
- [Derived] Asher L, Fekadu A, Teferra S, De Silva M, Pathare S, Hanlon C. "I cry every day and night, I have my son tied in chains": physical restraint of people with schizophrenia in community settings in Ethiopia. Global Health. 2017 Jul 11;13(1):47. doi: 10.1186/s12992-017-0273-1. PMID 28693614
- [Derived] Asher L, De Silva M, Hanlon C, Weiss HA, Birhane R, Ejigu DA, Medhin G, Patel V, Fekadu A. Community-based Rehabilitation Intervention for people with Schizophrenia in Ethiopia (RISE): study protocol for a cluster randomised controlled trial. Trials. 2016 Jun 24;17(1):299. doi: 10.1186/s13063-016-1427-9. PMID 27342215
- [Derived] De Silva MJ, Breuer E, Lee L, Asher L, Chowdhary N, Lund C, Patel V. Theory of Change: a theory-driven approach to enhance the Medical Research Council's framework for complex interventions. Trials. 2014 Jul 5;15:267. doi: 10.1186/1745-6215-15-267. PMID 24996765